CLINICAL TRIAL: NCT00440817
Title: A Review of Reports of Lymphoma Occurring in Patients With Rheumatoid Arthritis or Crohn's Disease in Centocor-Sponsored and Centocor-Supported Disease Registries
Brief Title: An Observational Study of Lymphoma in Patients With Rheumatoid Arthritis or Crohn's Disease.
Status: Completed | Type: Observational
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR011239; C0168T68 (Other: Centocor, Inc.)
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Lymphoma
Keywords: Lymphoma; Rheumatoid arthritis; Crohn's disease; Remicade; Infliximab
MeSH Terms: conditions — Lymphoma; Arthritis, Rheumatoid; Crohn Disease

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with lymphoma: Lymphoma Occurring in Patients with Rheumatoid Arthritis or Crohn's Disease
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — All treatments are prescribed by a physician on the basis of usual clinical practice.

SUMMARY:
The purpose of this study is to examine the association with EBV infection, monitor the occurrence of lymphoma and assess lymphoma risk in patients with rheumatoid arthritis and/or Crohns disease and you have taken infliximab.

DETAILED DESCRIPTION:
This is an observational (review of records), retrospective (research activity that is performed after the events under the study have occurred), registry study where data was collected from 3 different registries sponsored or supported by Centocor. Registries are Centocor-sponsored Therapy Resource Evaluation and Assessment Tool (TREAT™) Registry of Crohn's Disease, and in the following two Centocor-supported registries the Consortium of Rheumatology Researchers of North America, Inc. (CORRONA) registry and the Infliximab RA Registry, a subset of the National Database Registry of Rheumatoid Arthritis (NDBRRA) and of the National Databank for Rheumatic Diseases (NDB). A registry is data collection in a real life physician-patient setting. Physicians prescribe medications for rheumatoid arthritis and/or Crohns disease in accordance with their usual clinical practice and then record this information and provide it to Centocor. For this registry study, Centocor collected data from 3 registries to evaluate the risk of getting lymphoma if you have rheumatoid arthritis and/or Crohns disease and you have taken infliximab. Patients who were in one of the 3 registries and had rheumatoid arthritis and/or Crohns disease and did not take infliximab were also evaluated. This registry study does not involve the use of any investigational drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohns disease or rheumatoid arthritis who participate in the specified registries will be included in the analysis. For the lymphoma analysis, patients must be recorded as having a lymphoma during their participation in one of these registries

Exclusion Criteria:

* Patients who do not have Crohns disease or rheumatoid arthritis and who did not participate in one of the identified registries will be excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of lymphoma | 5 years
  To examine the occurrence of lymphoma among patients in one Centocor-sponsored and Centocor-supported disease registries

SECONDARY OUTCOMES:
Assessment of lymphoma risk | 5 years
  To assess lymphoma risk in relevant registry patient populations, including patients not receiving anti-TNF therapies, patients receiving conventional immunosuppressants (including corticosteroids), and patients receiving anti-TNF therapies
Evaluation of association of Epstein-Barr Virus (EBV) with the lymphoma | 5 years
  To evaluate all available data on tissue samples of individual lymphoma cases for the potential association of EBV with the lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Ortho Biotech Services, L.L.C. Clinical Trial, Study Director — Centocor Ortho Biotech Services, L.L.C.
Locations (3):
- United States (3):
  - Highland Park, Illinois
  - Wichita, Kansas
  - Albany, New York

REFERENCES:
- See also: A review of reports of lymphoma occuring in patients with rheumatoid arthritis or Crohn's disease in Centocor-sponsored or Centocor-supported disease registries. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=131&filename=CR011239_CSR.pdf